Barbed Suture: A Look at Its Use for Hysterotomy Closure During Cesarean Section

NCT04622267

PI: Calvin Lambert

Document Date: 8-15-2023

## 

Study ID: STUDY-20-01335 Form Version Date: 24MAR2023

## STUDY INFORMATION:

Study Title: Barbed Suture: A Look at its Use for Hysterotomy Closure During Cesarean Section

Study site: Icahn School of Medicine at Mount Sinai

**Principal Investigator (Lead Researcher):** Calvin E. Lambert, MD **Research Team:** Camila Cabrera, MD Clinical Fellow, MFM

Nicola Tavella, MPH Research Coordinator, MFM Nicola.tavella@mssm.edu

Physical Address: Mount Sinai OBGYN/MFM Faculty Practice Associates

5 E 98th St, 2nd Floor, New York, NY 10029

Mailing Address: One Gustave L Levy Place, Box 1171, NY, NY 10029

Phone: 646-823-7820

#### **SUMMARY OF THIS RESEARCH STUDY:**

This document explains a research study you might be interested in joining. Participation in the study is voluntary. You can agree to join or not. Your decision will not limit your ability to receive care at Mount Sinai. You should only agree to take part if you understand the study and if all of your questions about the research study are answered. If you do join the study, the research team must share any new information with you that may change your mind about taking part.

The purpose of this research study is to determine if barbed wire suture can decrease the amount of blood lost during a cesarean delivery, and if we can decrease the length of the procedure, as compared to using a vicryl suture. Barbed suture incorporates tiny barbs that distribute the tension along the entire suture line rather than the knotted ends as with traditional suture material. It is widely used in the field of minimally invasive gynecological surgery, however very few studies have looked at its use in obstetrics.

If you choose to take part, you will be asked to

- Deliver your baby at Mount Sinai Hospital (standard care).
- Be comfortable being randomized to either the barbed suture or traditional suture group.
- Allow study team to review your delivery record.
- Allow study team to contact you two weeks after your delivery discharge date to determine your pain level and if you developed any wound infection.

If you choose to take part, the main risks to you are a potential loss of confidentiality of your data. However, all efforts are made internally to preserve confidentiality of all data collected. You will not benefit directly from taking part in this research.

Instead of taking part in this research, you may opt to receive your physician's choice of suture.

If you are interested in learning more about this study, please continue to read below.

------FOR IRB USE ONLY-------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

| Study ID: STUDY-20-01335 | Form Version Date: 24MAR2023 |
|--------------------------|------------------------------|

#### STUDY PARTICIPATION:

You may qualify to take part in this research study because you are having a term, planned cesarean delivery at Mount Sinai Hospital.

Your participation in this research study is expected to last until completion of the two-week postpartum follow-up phone call.

There are 226 people expected to take part in this research study at Mount Sinai Hospital.

Funds for conducting this research study are provided by Icahn School of Medicine at Mount Sinai. Ethicon—the manufacturer, a subsidiary of Johnson & Johnson – are donating the suture material for this study.

## **DESCRIPTION OF WHAT IS INVOLVED:**

If you agree to take part in this research study, here is what may be involved:

- o Deliver your baby by c-section at Mount Sinai Hospital.
- The study treatment you get will be chosen by chance, like flipping a coin. Neither you nor the study doctor will choose what experimental study treatment you get. You will have an equal chance of being given the experimental treatment.
- Allow study team to review your medical records.
- Allow study team to contact you two weeks after your delivery discharge date to determine your pain level and if you developed any wound infection.

Because this research study involves the use of the Stratafix barbed suture, a note must be included in your electronic medical record that you are taking part in the research. This way, anyone involved in your medical care will know that you are a study participant, and they can work to avoid any problems or negative outcomes that could arise if they do not know.

#### Randomization

No one, not you, or anyone from your medical team or from the research team will be able to choose what group you are assigned to or what suture you get. It will be by chance, like flipping a coin. You will have an equal chance of being given each suture.

## **USE OF YOUR DATA AND/OR SAMPLES:**

The research team will never use or share your personal information (such as, name, address, date of birth, social security number), study data and/or samples (blood, tissue, urine, saliva, or any other body matter) that are collected as part of this study for future research, even if your identity is removed. Your data and/or samples will only be used to complete this study and then they will be destroyed.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

Study ID: STUDY-20-01335 Form Version Date: 24MAR2023

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for taking part in this study. Being in this study will not cost you anything extra.

#### **POSSIBLE BENEFITS:**

This study is not designed to benefit you personally. However, possible future benefits to others include improving clinical methods for cesarean delivery.

#### POSSIBLE RISKS AND DISCOMFORTS:

 Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

#### **OTHER OPTIONS TO CONSIDER:**

You may decide not to take part in this research study. If you decide not to take part, this will not affect the clinical care you receive at Mount Sinai. The choice is totally up to you.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY

If you believe that being in this research study has harmed you, you should contact the Lead Researcher. Their contact information is listed at the beginning of this consent form.

### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this study at any time. No matter what you choose, your care and benefits through Mount Sinai will not be negatively impacted.

If you decide to stop being in the study, please contact the Lead Researcher or the research staff.

You may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page. Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you decide you don't want your data and/or samples to be used for research anymore, you can contact the researcher and ask to have your data and/or samples withdrawn or labeled so that they

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

Form Version Date: 24MAR2023

Study ID: STUDY-20-01335

will not to be used in additional projects or shared. If your data and/or samples have already been shared with researchers, those researchers will be asked to stop using them. However, if any data and/or samples have already been shared without your identity or a linking code, it won't be possible to retrieve them. Data and/or samples that have already been used will not be affected by your decision. If your data and/or samples have already been deposited in an external repository, the study team will request that your data and/or samples be removed.

<u>Withdrawal without your consent</u>: The Lead Researcher, the funder or Mount Sinai may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the research team have not been followed, the Lead Researcher believes it is in your best interest, or for any other reason. If data and/or samples have been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT INFORMATION:**

If you have any questions, concerns or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Lead Researcher at phone number 646-823-7820

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Researchers sometimes get paid for consulting or doing work for companies that produce drugs, biologics or medical devices. If you have questions regarding industry relationships, you are encouraged to talk to the Lead Researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As part of this study, some of your private and/or protected health information will be obtained, used, and shared with your permission. There is a Federal Health Insurance Portability and Accountability Act (HIPAA) that makes sure this is done correctly and safely.

## What is protected health information (PHI)?

PHI is the combination of two things:

- 1. PHI contains information that identifies you. It will be used to contact you and link you to your health information, like name, date of birth, medical record number, and address.
- 2. PHI also contains health information, including information about your mental and physical health from your visits to doctors or hospitals, or from study visits.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

**Study ID: STUDY-20-01335** 

you are and your medical information.

Every time you visit a hospital or your doctor, PHI is created and recorded in your medical record by your healthcare providers. In the same way, the PHI created as part of this study will be linked to who

Form Version Date: 24MAR2023

What PHI is collected and used in this research study, and might also be shared with others? Gestational age, pregnancy outcomes, and pregnancy and obstetrical history

As part of this study, the research team at the hospital(s) involved in the research will collect your name, medical record number, telephone number, and dates directly related to you or your baby (birth date, admission date, discharge date).

During the study, the researchers will gather information by:

- Reviewing and/or taking your medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Completing the tests, procedures, questionnaires, and interviews explained in the description section of this consent.

#### Why is your PHI being used?

Researchers need the information that identifies you so they can contact you during the study. They need your health information and the results of any tests and procedures being collected as part of this study to answer the questions posed in the study. The purpose of the study is discussed earlier in this consent form. Before researchers analyze the data, they remove any information that would let others know who you are or that you took part in the study. If researchers publish or present study results at scientific meetings, lectures, or other events, their presentations would not include any information that would let others know who you are, unless you give separate permission to do so.

The Lead Researcher may also use and share the results of these tests and procedures with other healthcare providers at Mount Sinai who are involved in your care or treatment. The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example:

- The Mount Sinai Program for the Protection of Human Subjects is responsible for overseeing research on human participants and may need to see your information.
- If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes.
- If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

Who, outside Mount Sinai, might receive your PHI?

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

**Study ID: STUDY-20-01335** 

As part of the study, the Lead Researcher, research team and others in the Mount Sinai workforce may disclose your PHI, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Lead Researcher.)

 The United States Department of Health and Human Services (DHHS) and the Office of Human Research Protection (OHRP) (the government organization that is responsible for protecting human research participants).

Form Version Date: 24MAR2023

 A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.

In all disclosures outside of Mount Sinai, you will not be identified by any identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Lead Researcher will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board (IRB) allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, OHRP, as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

For how long will Mount Sinai be able to use or disclose your PHI? Your authorization for use of your PHI for this specific study does not expire.

#### Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The research team is not required to release research information to you that is not part of your medical record.

Do you need to give the researchers permission to obtain, use or share your PHI?

NO! If you decide not to let the research team obtain, use or share your PHI, you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment, or enrollment in any health plans or affect your eligibility for benefits.

#### Can you change your mind?

If you decide to stop being in the study, please contact the Lead Researcher or the research staff. The research team may ask you whether they can continue to collect information from your medical record. You will also have to decide if you wish to limit the continued use of the information collected

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

**Study ID: STUDY-20-01335** 

during the study. Under US privacy laws you may also withdraw your permission for the researchers to use and share any of your protected information for research, but you must do so in writing to the

Form Version Date: 24MAR2023

to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page.

Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected, but only to complete this research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your PHI.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If researchers are reviewing your medical records or asking questions about your medical history or conditions, it is possible that they may learn information related to your HIV status. If that is the case, the following information concerns you. If researchers are not reviewing your medical records or asking questions about your medical history or conditions, then you may ignore the following section.

#### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

## How the Institutional Review Board (IRB) can help you:

This research has been reviewed and approved by an Institutional Review Board (IRB). You may reach a representative of the Mount Sinai Program for Protection of Human Subjects at telephone number (212) 824-8200 during regular work hours (Monday-Friday, 9am-5pm, excluding holidays) for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 

Study ID: STUDY-20-01335 Form Version Date: 24MAR2023

| | our permission to take part in this rese<br>alth information. A signed and dated o | | |
|---|---|---|---|
| Signature of Participant | Printed Name of Participant | Date | Time |
| PERSON EXPLAINING STUDY A | ND OBTAINING CONSENT: | | |
| Signature of Consent Delegate | Printed Name of Consent Delegate | Date | Time |
| WITNESS SECTION: | | | |
| My signature below documents that the information in the consent document and any other written information was accurately explained to, and apparently understood by, the participant, and that consent was freely given by the participant. | | | |
| Signature of Witness | Printed Name of Witness | Date | Time |
| | FOR IRB USE ONLY | | |
| Rev 11.11.2022 (Amendment 1-03.09.2023 | | | |

IRB Approved